CLINICAL TRIAL: NCT02429752
Title: The Association of Breathing Pattern Dysfunction and Low Back Pain Presentation and Outcomes Following Physical Therapy
Brief Title: Low Back Pain and Breathing Pattern Dysfunction
Acronym: LBP&BPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Marlon Wong, Physical Therapist, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20140764
Record Dates: First submitted 2015-04-20; First posted 2015-04-29 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Low Back Pain
Keywords: inspiratory muscle training; low back pain; respiration; breathing
MeSH Terms: conditions — Low Back Pain; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inspiratory Muscle Training (Experimental): Subjects will receive 8 weeks of IMT
  Interventions: Other: Inspiratory muscle training

INTERVENTIONS:
Other: Inspiratory muscle training — Subjects that demonstrate unresolved BPD's upon reassessment after PT treatment, will have the option to participate in the second phase of the study. These subjects will be scheduled twice a week to receive IMT using the RT2 device and software program. The IMT protocol uses biofeedback to train at a specific percentage of MIP and SMIP for each inspiratory effort.

SUMMARY:
The goal of this study is to identify if there is a significant prevalence of abnormal respiratory patterns in a sample of patients with low back pain (LBP), and if the presence of abnormal respiratory patterns are predictive of rehabilitation outcomes in this population. In addition, the investigators will assess the response to inspiratory muscle training (IMT) for a subgroup of subjects that maintain abnormal breathing patterns after 1 month of physical therapy. Patients seeking physical therapy for LBP within the Uhealth system will be recruited. The first phase of this study will be observational. A comprehensive assessment of their respiratory function will be performed at the beginning of their therapy and after 1 month of therapy. Subjects that demonstrate abnormal respiratory patterns after 1 month of therapy will be offered the opportunity to participate in the second phase of the study in which they will receive 1 month of inspiratory muscle training (IMT). The respiratory assessment will then be repeated at the end of the IMT training program.

DETAILED DESCRIPTION:
The purpose of the first stage of this study is to assess the association and prognostic value of respiratory variables to low back pain presentation and outcomes with standard physical therapy care. Thus, a prospective longitudinal cohort, observational repeated measures (pre and post testing), design will be used for this portion of the study. Both the treating physical therapist and the patient will be blinded to the findings of the respiratory assessment in order to minimize the risk of treatment bias. Further, the physical therapy plan of care and the interventions administered will be at the therapists' discretion and will not be standardized. Typically a multimodal treatment approach is used for LBP, which includes: patient education, therapeutic exercises to improve strength, flexibility, and motor control deficits, manual therapy to decrease pain and improve joint and soft tissue mobility, and physical agents for pain management. By allowing therapists to use their clinical judgment, we are maintaining a real world environment which improves generalizability of the results. Although this will introduce variability that may confound results, there is no evidence that any single treatment approach is superior for addressing all LBP patients. Thus, allowing therapists to use their clinical reasoning to subgroup and treat accordingly maintains the standard of practice for all patient care.

A sample of convenience, consisting of 75 consecutive subjects seeking physical therapy for low back pain, will be selected. These subjects will be measured at the initiation of their physical therapy program and then retested 1 month later, using the procedures described below. Subjects with unresolved BPD's at the time of reassessment will be offered the opportunity to receive 1 month of inspiratory muscle training (IMT), which will be the second phase of this study. Subjects that complete the IMT will be retested following the same protocol at the end of the IMT program. All subject

recruitment and data collection will occur through UM facilities, but faculty at Nova Southeastern University will be involved with data analysis. Thus, IRB approval will be obtained from the University of Miami with a reliance agreement with Nova Southeastern University. It is anticipated that data collection will last from 6/2015-6/2016.

RESEARCH DESIGN AND METHODS

Subject recruitment

Patients seeking physical therapy for LBP at the University of Miami will be contacted by phone within 1 week of their initial examination. They will then be informed of the purpose of the study and the study protocol. If they express interest in participating, they will then be scheduled for a separate 90 minute session at the Kendall clinic during which all initial data will be collected. In addition, posters (see appendix 6) will be placed in the waiting room of 5 of the outpatient physical therapy clinics (Kendall, University of Miami Hospital, Bascom Palmer, Pain Center in CRB, and Plantation), all owned and operated by the University of Miami, as a recruitment tool as well. Qualifying patients from any of these facilities may call for additional information and to request inclusion in the study as well.

Measurement protocol

Resting Baseline Data

First subjects will be interviewed to collect data on their condition and status, as well as to screen for inclusion/exclusion criteria. (see Appendix 1 for data collection sheet). The subjects will then be asked to complete 3 questionnaires: the Pain Catastrophizing Scale, the Modified Oswestry Disability Index, and the Nijmegen Questionnaire (Appendix 2, 3, and 4 respectively). These questionnaires should take less than 5 minutes each to complete. Prior to beginning physical data collection, subjects will be informed to immediately stop any activity that causes significant discomfort or increased symptoms during the testing session. Then, subjects will be asked to breath forcefully into the Micro MPM (Micro Medical Ltd, Chatham, UK) device in order to collect MEP. This will be repeated 3-5 times with a 1 minute rest in between each trial. They will then be asked to place the TIRE device in their mouth and breathe in forcefully and sustain the breath for as long as possible in order to collect MIP and SMIP data. This process will also be repeated 3-5 times. Finally, the subjects will be fitted with the Cosmed K4b2 and Respitrace systems; these devices will be described in detail later. The k4b2 consists of a rubber mask with a light nylon vest to measure breath by breath gas analysis, and the Respitrace consists of merely 2 soft chest straps to measure heart rate variability and chest excursion with breathing. The subjects will then lie in the supine position for 5 minutes, sit quietly for 5 minutes, and stand quietly for 5 minutes in order to gather baseline data in each of these positions. The first 2 minutes in each position will be used as an accommodation period and data will not be recorded. Thus data analysis will only consist of the data from the final 3 minutes in each of these positions.

Postural Challenge baseline data

Subjects will be seated in a stable chair, with the feet on the ground and without back support, and asked to perform 3 rounds of resisted shoulder flexion and resisted hip flexion on each extremity. A submaximal resistance will be applied manually by the investigator and held for 30 seconds followed by 30 seconds of rest. After, they will be asked to lift and hold a 25 lb weight for 30 seconds 3 times, followed by 30 seconds of rest between each trial. Then they will lift the weight 10 times repetitively in a faster paced rhythmic fashion set by a metronome. They will then rest in the seated position for 5 minutes to measure recovery heart rate and respiration.

Inspiratory Muscle Training (IMT)

Subjects that demonstrate unresolved BPD's upon reassessment after PT treatment, will have the option to participate in the second phase of the study. These subjects will be scheduled twice a week to receive IMT using the RT2 device and software program (described in detail later). The IMT protocol uses biofeedback to train at a specific percentage of MIP and SMIP for each inspiratory effort. The program consists of 6 breaths per level, with 6 levels, and the ability to alter the rest time between breaths as the subject advances through each of the levels. The training session is completed when the subject fails to achieve the selected percentage of SMIP twice consecutively, or if they complete all 6 levels for a maximum of 36 breaths. The IMT program will be set at 60% of each subjects MIP/SMIP and breathing at this workload will focus on full deep inhalations using diaphragmatic breathing followed by slow prolonged exhalations with each subsequent inhalation being signaled by the RT2 software prompt (via visual display on the computer screen) to "Please Inhale". The first level of IMT will consist of a 40 second rest period between breaths followed by a 30 and 20 second rest period during IMT at levels 2 and 3, respectively. The rest period during IMT at the remaining three levels will remain at 20 seconds during which subjects will be prompted to prolonged exhalation throughout as much of the 20 second rest period as possible. The training session will also be stopped if the subject complains of increased back pain and if dizziness, fatigue, or if any other adverse response is noted.

Post IMT Data Collection

After 4 weeks, or 8 sessions of IMT, the same data collection protocol will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65,
* seeking physical therapy services for lumbar or pelvic pain will be recruited for this study.
* Subjects must intend to complete their prescribed physical therapy plan of care.

Exclusion Criteria:

* Patients unable to consent, complete questionnaires independently, or fulfill all testing requirements will be excluded from the study.
* All vulnerable populations will be excluded including:

  * prisoners,
  * children,
  * terminally ill patients, and
  * individuals with cognitive, emotional, or communication impairments that require them to have a guardian.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in baseline value of breath-by-breath gas analysis | baseline, after 1 month of therapy, after 2 months of IMT
  Measure of breathing pattern and respiratory gases at rest and with activity

SECONDARY OUTCOMES:
Number of Participants improved on the Oswestry Disability Index | baseline, after 1 month of therapy, after 2 months of IMT
  The modified Oswestry Disability Index (ODI), also referred to as the Low Back Disability Questionnaire, is an anatomic region based questionnaire used to assess self-report disability (Appendix 3). The ODI is a 10 item questionnaire with each item scored on a 6 point scale (0-5). Total scores can range from 0-50 with higher scores representing more disability. Scores are then converted into a percentage with 0-20% representing minimal disability, 20-40% moderate disability, 40-60% severe disability, 61-80% crippled, and 80-100% as bed-bound or symptom magnification.
Number of Participants improved on the Numeric Pain Rating Scale | baseline, after 1 month of therapy, after 2 months of IMT
  The Numeric Pain Rating Scale (NPRS) is an 11 point scale from 0-10, with 0 representing "no pain" and 10 representing "the worst pain imaginable"
Change in baseline value of Maximal inspiratory pressure | baseline, after 1 month of therapy, after 2 months
  Test of respiratory muscle strength
Change in baseline value of sustained maximal inspiratory pressure | baseline, after 1 month of therapy, after 2 months
  Test of respiratory muscle strength
Change in baseline value of maximal expiratory pressure | baseline, after 1 month of therapy, after 2 months
  Test of respiratory muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Marlon L Wong, DPT, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States